CLINICAL TRIAL: NCT06300697
Title: Michigan Food and Atopic Dermatitis (M-FAD) Program - Molecular Analytics Project
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Charles (Chase) Schuler, Assistant Professor of Internal Medicine and Assistant Professor of Mary H Weiser Food Allergy, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00235532
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis; Food Allergy; Healthy
Keywords: Blood Samples; Skin Samples; Transepidermal water loss (TEWL) monitor; Allergic reaction
MeSH Terms: conditions — Dermatitis, Atopic; Food Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control group Adult (Other): Participation will be approximately 14 days after enrollment.
  Interventions: Other: Data and biospecimen collection; Other: Skin biopsies; Other: Oral Food Challenge (OFC) procedures
- Food allergy-only group (Other): Participation will be approximately 14 days after enrollment.
  Interventions: Other: Data and biospecimen collection; Other: Skin biopsies; Other: Oral Food Challenge (OFC) procedures
- Food allergy plus atopic dermatitis group (Other): Participation will be approximately 14 days after enrollment.
  Interventions: Other: Data and biospecimen collection; Other: Skin biopsies; Other: Oral Food Challenge (OFC) procedures
- Atopic dermatitis without food allergy group (Other): Participation will be approximately 14 days after enrollment.
  Interventions: Other: Data and biospecimen collection; Other: Skin biopsies; Other: Oral Food Challenge (OFC) procedures
- Control Group less than 18 years old (Other): Participation will be approximately 14 days after enrollment.
  Interventions: Other: Data and biospecimen collection; Other: Oral Food Challenge (OFC) procedures

INTERVENTIONS:
Other: Data and biospecimen collection — Enrolled participants will have health-related information and blood specimens collected.
Other: Skin biopsies — Participants will be asked to provide one or two skin biopsies (days 1 and 2) from the forearm, unless the participant is a healthy child (no food allergy and no atopic dermatitis), in which case there will be no skin biopsy.
  Arms: Atopic dermatitis without food allergy group; Control group Adult; Food allergy plus atopic dermatitis group; Food allergy-only group
Other: Oral Food Challenge (OFC) procedures — Participants will have the choice of consenting to an OFC (approximately 2-4 hours) to peanut, tree nut, egg, milk, or sesame. If there is no allergy history, the study team will conduct an oral food challenge to one of the choices. The OFC will occur in the clinical research area. and done the same as a clinical care OFC. A transepidermal water loss monitor will be applied to participant's arm with a sticky pad and will stay on the arm for the challenge. Food doses will be given in small amounts that increase in size up to a defined single serving of the food based upon the participants age/size. The OFC will proceed until a full dose is consumed without symptoms, or until anaphylaxis occurs. Depending upon the participant's reaction to the oral food challenge, the participant may be requested to return the next day for a research visit that would take less than an hour. The 24-hour post oral food challenge visit will include an interview to assess condition and a blood sample.

SUMMARY:
This study will explore potential links between atopic dermatitis and food allergy. This information will be useful to determine atopic dermatitis and food allergy share unique biochemical or genetic identifiers useful for diagnosing and treatments in the future.

This is a mechanistic study consisting of obtaining blood and skin samples from participants at baseline. Individuals may also undergo a clinically indicated oral food challenge and have blood and skin samples collected at various times during the oral food challenge. This study will create a molecular map of the pathology of atopic dermatitis and food allergy. This information will be deployed to evaluate the hypothesis that atopic dermatitis and food allergy share unique genetic transcriptional signals in which the study team can then further analyze pathological pathways and cell types.

DETAILED DESCRIPTION:
This study will be funded by the National Institute of Health. Once the funds are received, the registration will be updated with this information.

ELIGIBILITY:
Food allergy-only group Inclusion Criteria:

* Have a known history of food anaphylaxis to peanut, tree nut, egg, milk, or sesame confirmed by an allergist.
* Have had skin and blood food allergy testing to the food allergen in question within the past 6 months. Meet the 80% likelihood positive predictive value threshold for allergy based on at least 1 of either the skin or blood immunoglobulin E (IgE) tests per current literature corrected for age. See protocol for more details.
* No history of atopic dermatitis

Food allergy plus atopic dermatitis group Inclusion Criteria:

- Meet the "food allergy only group" inclusion criteria except this group must also have atopic dermatitis.

Atopic dermatitis without food allergy Inclusion Criteria:

* Have a present diagnosis of atopic dermatitis by an allergist and/or dermatologist.
* Have no history of food allergy, past or present.

Control Group Inclusion Criteria:

- No history of food allergy or atopic dermatitis, past or present.

Exclusion Criteria for all groups:

* People younger than age 10 or older than age 55
* Any active cardiovascular disease, cancer, pulmonary disease except well-controlled asthma, or other condition that would preclude an OFC otherwise. Mild conditions that would not preclude an OFC are allowed (i.e., controlled hypertension or a surgically removed skin cancer that is resolved would not be exclusionary for this study, for example).
* Any medication use that cannot be stopped temporarily for the OFC that would interfere with the OFC result. Medications in this category include antihistamines (first or second generation) within 1 week.
* Any skin condition aside from atopic dermatitis per inclusion criteria groups that might impact the study, including such conditions as autoimmune skin conditions (such as psoriasis), congenital ichthyoses, hyper-IgE syndromes.
* Any recent change (within 6 months) of starting or stopping a biologic medication, such as dupilumab, tezepelumab, or others that might interfere with atopic dermatitis or food allergy.
* Any past or present history of oral immunotherapy (OIT) for any food allergen.
* Pregnancy - females of childbearing age will be asked and self-report pregnancy status.

Ages: 10 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Anaphylaxis occurrence rates in each group | Approximately 4 hours (Day 1 during the food challenge)
  Anaphylaxis likelihood will be defined by the Brighton criteria. Any Brighton Level 1, 2, or 3 anaphylaxis. Score 1 = definite anaphylaxis, score 2 = probable anaphylaxis, score 3 = possible anaphylaxis.

SECONDARY OUTCOMES:
Anaphylaxis severity in each group | Approximately 4 hours (Day 1 during the food challenge)
  This will be graded on a scale of 1 to 5 (where 1 = mild, 5 = death) according to criteria set forth in the Consortium for Food Allergy Research (CoFAR) Grading Scale.
Reaction rates in each group | Approximately 4 hours (Day 1 during the food challenge)
  Any objective symptom of allergic reaction occurs (e.g., hives, angioedema, vomiting, wheeze, etc.) not rising to the definition of anaphylaxis.
Anaphylaxis likelihood in each group based on the Brighton score | Approximately 4 hours (Day 1 during the food challenge)
  The Brighton score gives a 0-3 score of anaphylaxis likelihood (0 = no anaphylaxis, 3 = highly likely).

CONTACTS AND LOCATIONS:
Overall Officials: Chase Schuler, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No